CLINICAL TRIAL: NCT03340441
Title: Clinical Evaluation for Body Temperature Measurement Using Prizma Smart Phone Cover and Application
Brief Title: Prizma Device Temperature Measurement
Acronym: Prizma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: G Medical Innovations Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-7.4.7.10.10
Record Dates: First submitted 2017-10-24; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Prizma — sensor unit with mobile application installed on smartphone
  Other Names: Smartphone cover / Jacket

SUMMARY:
The purpose of the study is to evaluate the temperature measurements by the Prizma device.

DETAILED DESCRIPTION:
Primary objective of this study is to compare the temperature measured by the PRIZMA to the oral and Armpit temperature measured by a gold standard device in order to develop and evaluate a skin to body temperature conversion table.

Secondary objective is to collect and compare data of ECG, Respiration and SpO2 collected from the Prizma device to the data collected from gold standard devices for reference of noise level and for future development of the PRIZMA device.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age above 18 years from both genders
* ASA physical status 1-4
* Hospitalized in internal ward

Exclusion Criteria:

* Abuse of alcohol or illicit drugs
* History of mental retardation or any mental disease
* Skin irritation / Atopic dermatitis or any other skin condition at the area of patients palms that might affect his/her ability to hold the device appropriately

Ages: 17 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalised adults of which the total number of febrile subjects shall not be less the 30% and not greater than 50% of all subjects.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Temperature measurement | 3 months
  Develop and evaluate a skin to body temperature conversion table.

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Tishler, Prof., Principal Investigator — Asaf Harofe Medical Center
Locations (1):
- Asaf Harofe Medical Center, Rishon LeZiyyon, Israel

IPD SHARING:
Plan to Share IPD: No